CLINICAL TRIAL: NCT06621836
Title: Analgesic Efficacy of Intermediate Cervical Plexus Block in Patients Undergoing Neck Surgeries: A Comparison Between Two Bupivacaine Concentrations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-425-2023
Record Dates: First submitted 2024-07-12; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Cervical Plexus Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-H (Active Comparator)
  Interventions: Drug: ICPB H
- Group-L (Active Comparator)
  Interventions: Drug: ICPB - L

INTERVENTIONS:
Drug: ICPB H — ICPB technique The patient's head will be rested on a pillow and turned to the opposite side. A linear probe with higher frequencies will be placed transversely over the midpoint of the SCM muscle. The carotid artery will be identified and traced upwards to its bifurcation. the probe will be then moved laterally to identify the tapering posterolateral end of the SCM muscle. Via an in-plane technique, a 22-gauge, 50 mm needle will be advanced underneath the investing fascia of SCM muscle and above the interscalene groove until feeling the "pop" on piercing the investing fascia. The patient will be then randomly allocated into two groups (H & L) using computer-generated random numbers that will be concealed in opaque envelopes. Group H will receive 10 ml 0.25 % bupivacaine he technique will be repeated on the opposite side
  Arms: Group-H
Drug: ICPB - L — ICPB technique The patient's head will be rested on a pillow and turned to the opposite side. A linear probe with higher frequencies will be placed transversely over the midpoint of the SCM muscle. The carotid artery will be identified and traced upwards to its bifurcation. the probe will be then moved laterally to identify the tapering posterolateral end of the SCM muscle. Via an in-plane technique, a 22-gauge, 50 mm needle will be advanced underneath the investing fascia of SCM muscle and above the interscalene groove until feeling the "pop" on piercing the investing fascia. The patient will be then randomly allocated into two groups (H & L) using computer-generated random numbers that will be concealed in opaque envelopes. Group L will receive 10 ml 0.125% bupivacaine. The technique will be repeated on the opposite side
  Arms: Group-L

SUMMARY:
Cervical plexus blocks (CPB) have been widely used to provide effective anesthesia and analgesia during various head and neck procedures. The ICPB was considered a good alternative to the deep CPB with an easier technique and fewer adverse events such as intravascular, epidural, subarachnoid injection, and phrenic nerve palsy. A recent randomized trial investigated the analgesic efficacy of superficial vs intermediate CPB combined with GA during total thyroidectomy. Authors used 10 ml bupivacaine 0.25% bilaterally, and they revealed a lower pain score and prolonged duration of analgesia with ICPB compared to superficial CPB; however, the authors did not assess the influence of this bupivacaine concentration on the diaphragmatic motion. [5] This randomized comparative trial is designed to investigate the analgesic efficacy of ICPB combined GA using two bupivacaine concentrations in patients undergoing neck surgeries (total thyroidectomy or total laryngectomy). We hypothesize that a smaller concentration of bupivacaine (0.185%) could provide an equivalent analgesic effect to a larger concentration (0.25%) with less impact on the diaphragmatic motion. The primary endpoint is the duration of postoperative analgesia. The secondary endpoints are the intraoperative hemodynamics, the postoperative pain score, total postoperative opioid consumption over 24 hours, diaphragmatic motions, and hemi-diaphragmic paresis.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III,
* scheduled for total thyroidectomy or total laryngectomy

Exclusion Criteria:

* Heart failure,
* A history of arrhythmias or treatment with antiarrhythmic drugs,
* Impaired pulmonary, liver or kidney functions,
* Neck infection or rash

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
The duration of analgesia | Time elapsed from the end of the ICPB block procedure till VAS ≥ 4 over 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia department - Faculty of medicine- Cairo University, Cairo, Egypt